CLINICAL TRIAL: NCT02821585
Title: Impact of a Nutritional Intervention on Type1 Diabetes Adult With Metabolic Syndrome
Acronym: MEDIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEDIT-1
Record Dates: First submitted 2016-06-20; First posted 2016-07-01 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2017-09

CONDITIONS: Type 1 Diabetes; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Metabolic Syndrome | interventions — Nutrition Assessment

ARMS (2):
- Mediterranean Diet (Active Comparator): Participants will receive nutritional lessons on the principles of the Mediterranean diet. This type of diet is defined with a carbohydrate intake of 45-55% of total energy intake, 15-20% of proteins, 30-35% of lipids and less than 7% for saturated fat. Nine sessions with a nutritionist are planned to cover various topics of the diet.
  Interventions: Behavioral: Nutritional Counseling
- Low Fat Diet (Placebo Comparator): Participants will receive nutritional lessons on the principles of the low fat diet. This type of diet is defined with a carbohydrate intake greater than 45% of total energy intake, 15-20% of proteins, less than 30% of lipids and less than 7% for saturated fat. Nine sessions with a nutritionist are planned to cover various topics of the diet.
  Interventions: Behavioral: Nutritional Counseling

INTERVENTIONS:
Behavioral: Nutritional Counseling — Carbohydrate counting will be reviewed, as well as hypoglycemia management. The 9 following visits will focus on different aspects of each diets: types of fats, meat and alternatives, grain products, milk and alternatives, fruits and vegetables, salt intake, energy density and restaurants.

SUMMARY:
Recent studies have found that up to 45 % of patients with type 1 diabetes have metabolic syndrome, a cluster of conditions (abdominal obesity, hypertension, dyslipidemia, insulin resistance) that increase the cardiovascular risk. The investigators have observed in previous studies a strong association between the adherence to a Mediterranean diet and the prevalence of metabolic syndrome on patients with metabolic syndrome. However, no intervention has been realized on this population and the current recommendations (low fat diet) differ from the Mediterranean diet. A nutritional intervention on the principles of the Mediterranean diet could therefore play a role in the treatment of the metabolic syndrome in Type 1 diabetes patients. The main objective of this study is to examine the impact of a nutritional intervention on the waist circumference after 6 months of an intervention group (Mediterranean diet) versus a control group (low fat diet).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes for at least 12 months
* On intensive insulin therapy with multiple daily injections or on insulin pump
* Be overweight or obese (BMI≥25 kg/m2)
* Stable weight for at least 3 months
* If on medication for thyroid, hypertension or dislipidemia: stable doses in the last 3 months
* Presenting at least 3 of the 5 following criteria for metabolic syndrome:

  1. Waist circumference >102cm ♂ or >88cm ♀
  2. Triglycerides >1.7mmol/L or medication
  3. Cholesterol-HDL <1.0mmol/L ♂ or <1.3mmol/L ♀ or medication
  4. Blood pressure ≥130/85 mmHg or medication
  5. Estimated insulin resistance (eGDR <6.29)

Exclusion Criteria:

* Mental incapacity, refusal or linguistic barrier that could affect comprehension or cooperation with the study
* Ongoing pregnancy
* Diet corresponding to the criteria of a mediterranean diet (score≥27)
* Vegetarianism
* Major diabetes complications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change in Waist Circumference | Change from baseline and 6 months measure of waist circumference
  The outcome will be measured every month, at admission and visits 4 (1 month) - 6 (2 months) -7 (3 months) -8 (4 months) -9 (5 months) -10 (6 months) -11 (9 months).

SECONDARY OUTCOMES:
Mediterranean Diet Score | The outcome will be measured based on an internet food frequency questionnaire filled by patients at admission, visit 7 (3 months) and visit 10 (6 months).
  The questionnaire allows the calculation of a score reflecting the adherence to the mediterranean diet.
Body Mass Index (BMI) | Weight wil be measured every month: at admission and visit 4 (1 month), 6 (2 months), 7 (3 months), 8 (4 months), 9 (5 months) and 10 (6 months). The height will be measured only at admission.
  Weight (kg) / (height (m) x height (m))
Percentage of body fat | The outcome will be measured at admission, visit 7 (3 months) and visit 10 (6 months)
  The outcome will be measured using a DEXA-scan
Insulin Sensitivity | The outcome will be calculated at admission, visit 7 (3 months) and visit 10 (6 months)
  The outcome will be estimated based on a formula validated for type 1 diabetes subjects. The formula takes into account waist/hip ratio, glycated hemoglobin and hypertension.
Systolic and diastolic Blood pressure | The outcome will be measured at admission, visit 7 (3 months) and visit 10 (6 months)
  Average of 3 measures (systolic, diastolic and pulse) after a 5 minutes resting period
Lipid profile | The outcome will be measured at admission, visit 7 (3 months) and visit 10 (6 months)
  A blood test will measure level of total cholesterol, triglycerides and LDL cholesterol.
Glycemic variability | The outcome will be measured at admission, visit 7 (3 months) and visit 10 (6 months)
  Glycated hemoglobin will be measured with a blood sample. Hypoglycemia frequency will be measured with a 4-day glycemia journal.

CONTACTS AND LOCATIONS:
Overall Officials: Remi Rabasa-Lhoret, Study Director — IRCM
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Fortin A, Rabasa-Lhoret R, Lemieux S, Labonte ME, Gingras V. Comparison of a Mediterranean to a low-fat diet intervention in adults with type 1 diabetes and metabolic syndrome: A 6-month randomized trial. Nutr Metab Cardiovasc Dis. 2018 Dec;28(12):1275-1284. doi: 10.1016/j.numecd.2018.08.005. Epub 2018 Aug 30. PMID 30459054